CLINICAL TRIAL: NCT00998699
Title: A Randomized, Double-blind, Placebo-controlled, Phase 2 Study of the Effects of XOMA 052 on Insulin Production in Subjects With Well-controlled Type 1 Diabetes
Brief Title: Study of the Effects of XOMA 052 on Insulin Production in Subjects With Well Controlled Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: X052076
Record Dates: First submitted 2009-10-19; First posted 2009-10-20 (Estimated); Last update posted 2014-03-04 (Estimated); Status verified 2014-03

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — gevokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- XOMA 052 (Active Comparator)
  Interventions: Drug: Xoma 052
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Xoma 052 — Sterile solution subcutaneously administered every 4 weeks for 12 weeks
  Arms: XOMA 052
Drug: Placebo — Sterile solution subcutaneously administered every 4 weeks for 12 weeks
  Arms: Placebo

SUMMARY:
The study hypothesis is that XOMA 052 may inhibit beta-cell destruction and enhance beta-cell regeneration.

The purpose of this study is to assess the effects of XOMA 052 on beta-cell function and insulin production.

ELIGIBILITY:
Inclusion criteria:

* Stable Type 1 diabetes of > 2 year duration
* No clinically significant change in treatment regimen for T1D
* Age ≥ 18 years and ≤ 55 years
* HbA1c < 7.0%
* Positive GAD65 and/or IA-2 auto-antibodies
* Peak C-peptide > 100 pM following IV injection of 1 mg glucagon
* Body-mass index (BMI) > 18 and < 28 kg/m2
* Willingness to maintain current doses/regimens of vitamins and dietary supplements through the end of the study

Exclusion criteria:

* Current infection or history of infection
* Positive for Hep B surface antigen (HBsAg), Hep C virus (HCV), or HIV
* History of tuberculosis or positive PPD test
* Presence of foot, leg, or decubitus ulcers
* Current immunosuppressive treatment or documented immunodeficiency
* History of severe allergic or anaphylactic reactions
* History of asthma requiring systemic corticosteroid therapy
* Coronary intervention (PCI, stent placement) or hospitalization for cardiovascular condition within the last 12 months
* Uncontrolled hypertension
* History of congestive heart failure (NYHA Class III or IV)
* History of a coronary event within the last 12 months
* Female subjects who are pregnant, planning to become pregnant, have recently delivered, or are breast-feeding
* History of malignancy within the last 5 years
* Receipt of a live (attenuated) vaccine within the last 3 months

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-02; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in beta-cell function as measured by change in C-peptide level during thd MMTT (Mixed meal tolerance test) at Day 112 compared to baseline (Day 0 pre-dose) | Day 0 pre-dose and Day 112

SECONDARY OUTCOMES:
Safety assessed by pre- and post-treatment serial measurements of vital signs, clinical laboratory assessments, and treatment-emergent adverse events. | Day 0 (baseline) through Day 364
Change in insulin requirements | Day -3 through Day 0 pre-dose and Day 109 through Day 112)
Change in HbA1c levels | Day 0 pre-dose and Day 112
Change in fasting glucose | Day 0 pre-dose and Day 112
Change in fasting glucagon and cortisol | Day 0 pre-dose and Day 112
Change in systemic inflammation markers | Day 0 pre-dose and Day 112
Change in meal-stimulated GLP-1 and GIP | Day 0 pre-dose and Day 112
Change in lipids profile | Day 0 pre-dose and Day 112
Measurement of serum concentrations of XOMA 052 | Day 0 pre-dose, Day 28, Day 56, Day 84, Day 112, Day 182, and Day 364

CONTACTS AND LOCATIONS:
Overall Officials: Marc Donath, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (2):
- Switzerland (2):
  - Basel
  - Zurich